CLINICAL TRIAL: NCT05479799
Title: Prevalence and Determinants of Anemia During the Third Trimester of Pregnancy
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel-Tawab Mahmoud, MD, Principal Investigator, Beni-Suef University
Other Study IDs: anemia in pregnancy: Beni-Suef
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Anemia of Pregnancy
Keywords: Anemia; Hemoglobin; Third trimester; Pregnancy outcome
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anemia group: anemia was diagnosed with a hemoglobin level of less than 11.0 g/dl
- Non-anemia group: Normal hemoglobin was diagnosed with a hemoglobin level of more than 11.0 g/dl

SUMMARY:
This cross-sectional study was conducted on 383 pregnant women who attended the antenatal care clinic during their third trimester at Beni-Suef University Hospital.

A proper history was taken from each participant. All women were subjected to routine antenatal care, including physical examinations, ultrasound examinations, and routine laboratory tests.

According to WHO criteria, anemia was diagnosed with a hemoglobin level of less than 11.0 g/dl. Anemia was further divided into three degrees; mild with hemoglobin level 10-10.9 g/dl, moderate with hemoglobin level 7-9.9 g/dl, and severe with hemoglobin level < 7.0 g/dl.

DETAILED DESCRIPTION:
This cross-sectional study was conducted on 383 pregnant women who attended the antenatal care clinic during their third trimester at Beni-Suef University Hospital.

A proper history was taken from each participant regarding age, educational level, residency (urban or rural), occupation, family income, frequency of antenatal visits, obstetric history, medical history, and surgical history. Nutritional history is taken to detect the frequency intake of meat/month, chicken/week, fish/week, fruits/week, vegetables/week, and tea/day. History of iron supplements intake was taken. All women were subjected to routine antenatal care, including a physical examination (e.g., measuring blood pressure), ultrasound, and umbilical artery Doppler examination. A blood sample was taken from each enrolled woman for standard laboratory tests such as complete blood picture, blood group, RH type, and blood sugar test if there is a risk. A urine sample was taken for urine analysis. Blood from each participant was drawn from the cubital vein into appropriate blood collection tubes using vacuum tube needles (Becton Dickinson Medical Devices Co. Ltd., Franklin Lakes, USA). K2EDTA tubes were used for CBC. Samples were transported and tested within 4 hours after collection. Measured CBC parameters included RBC, HGB, HCT, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), MCH concentration (MCHC), platelet count (PLT), WBC, and WBC differentials, including percentages and absolute counts of neutrophils (NEUT% and NEUT), lymphocytes (LYM% and LYM), monocytes (MONO% and MONO), basophils (BASO% and BASO), and eosinophils (EO% and EO).

According to WHO criteria, anemia was diagnosed with a hemoglobin level of less than 11.0 g/dl. Anemia was further divided into three degrees; mild with hemoglobin level 10-10.9 g/dl, moderate with hemoglobin level 7-9.9 g/dl, and severe with hemoglobin level < 7.0 g/dl.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women during their third trimester

Exclusion Criteria:

* Women with chronic medical illness

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included pregnant women who attended the antenatal care clinic during their third trimester.
Sampling Method: Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with the prevalence of anemia in the third trimester of pregnancy | through study completion (3-6 months)
  Number of participants with the prevalence of anemia in the third trimester of pregnancy in a specific geographical area (Beni-Suef University Hospital as a tertiary referral center)

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Banī Suwayf, Egypt